CLINICAL TRIAL: NCT07028710
Title: Evolution of Luteal Progesteronemia in a Modified Natural Cycle (Ovulation Triggered by hCG): Pilot Study
Brief Title: Early Luteal Phase Progesterone Kinetics After hCG-Induced Ovulation in Modified Natural Cycle
Acronym: CineP4
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: RECHMPL24_0200
Record Dates: First submitted 2025-06-11; First posted 2025-06-19 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Luteal Phase Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: hCG

INTERVENTIONS:
Drug: hCG — Subcutaneous injection of 250 µg of recombinant hCG (Ovitrelle®)

SUMMARY:
This pilot study evaluates how progesterone levels change after hCG-triggered ovulation in modified natural cycles. Forty women preparing for frozen embryo transfer will have blood tests over 6 days to monitor hormone levels. The goal is to understand whether hCG affects the timing of the luteal phase and embryo implantation.

ELIGIBILITY:
Inclusion Criteria:

* At least 1 follicle of 17 mm or more
* Endometrium of 6 mm or more
* Plasma luteinizing hormone (LH) less than 2 times basal level (measured at the beginning of the cycle between D1 and D4) and progesteronemia less than 1.5 ng/mL
* For whom ovulation induction with recombinant hCG (Ovitrelle) is then proposed (standard care).

care)

Exclusion Criteria:

* Patient whose venous capital contraindicates repeated blood sampling over a short period of time over a short period.
* Patient treated with exogenous natural progesterone (vaginal or injectable) which may interfere or synthetic progesterone, which may interfere with endogenous progesterone secretion.
* Patient who has not given written consent to participate in the study.
* Patient not fluent in French.
* Patient under guardianship, curators or without social security coverage.
* Patient participating in another study with an ongoing exclusion period or other interventional research with no ongoing exclusion period involves the use of a drug or procedure capable of altering progesterone levels .

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Enrollment: 40 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2028-06-15 (Estimated); Study Completion 2030-06-15 (Estimated)

PRIMARY OUTCOMES:
Serum Progesterone Level on Day 3 After hCG Trigger | 3 Days After hCG Injection

CONTACTS AND LOCATIONS:
Overall Officials: Noémie RANISAVLJEVIC, Investigator Coordinator, Principal Investigator — CHU de Montpellier

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mizrachi Y, Horowitz E, Ganer Herman H, Farhi J, Raziel A, Weissman A. Should women receive luteal support following natural cycle frozen embryo transfer? A systematic review and meta-analysis. Hum Reprod Update. 2021 Jun 22;27(4):643-650. doi: 10.1093/humupd/dmab011. PMID 33829269
- [Background] Lee VC, Li RH, Chai J, Yeung TW, Yeung WS, Ho PC, Ng EH. Effect of preovulatory progesterone elevation and duration of progesterone elevation on the pregnancy rate of frozen-thawed embryo transfer in natural cycles. Fertil Steril. 2014 May;101(5):1288-93. doi: 10.1016/j.fertnstert.2014.01.040. Epub 2014 Mar 3. PMID 24602752
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/24602752/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/32395750/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/33829269/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/27798046/